CLINICAL TRIAL: NCT05152459
Title: A Phase 1/2 Study of Tazemetostat With Umbralisib and Ublituximab in Patients With Relapsed/Refractory Follicular Lymphoma
Brief Title: Tazemetostat in Combination With Umbralisib and Ublituximab for the Treatment Relapsed or Refractory Follicular Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Feasibility
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21303; NCI-2021-12560 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21303 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Follicular Lymphoma; Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tazemetostat; ublituximab; LFB-R603; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tazemetostat, umbralisib, ublituximab) (Experimental): Patients receive ublituximab IV on days 1, 8, and 15 of cycle 1, day 1 of cycle 2-6, and day 1 of every 3 cycles thereafter. Patients also receive tazemetostat PO BID umbralisib by PO QD on days 1-28. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tazemetostat; Biological: Ublituximab; Drug: Umbralisib

INTERVENTIONS:
Drug: Tazemetostat — Given PO
  Other Names: E7438; EPZ-6438; EPZ6438
Biological: Ublituximab — Given IV
  Other Names: LFB-R603; TG-1101; TG-20; TGTX-1101
Drug: Umbralisib — Given PO
  Other Names: 2-((1S)-1-(4-Amino-3-(3-fluoro-4-(1-methylethoxy)phenyl)-1H-pyrazolo(3,4-d)pyrimidin-1-yl)ethyl)-6-fluoro-3-(3-fluorophenyl)-4H-1-benzopyran-4-one; RP-5264; RP5264; TGR-1202

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose of tazemetostat and umbralisib and whether tazemetostat in combination with umbralisib and ublituximab works to shrink tumors in patients with follicular lymphoma that has come back (relapsed) or does not respond to treatment (refractor). Tazemetostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Umbralisib may help block the formation of growths that may become cancer. Ublituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving tazemetostat in combination with umbralisib and ublituximab may work better in treating follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of a regimen combining tazemetostat, umbralisib and ublituximab in patients with relapsed/refractory follicular lymphoma (FL).

II. Estimate the overall response rate (ORR) in relapsed/refractory FL patients treated with tazemetostat, umbralisib and ublituximab.

SECONDARY OBJECTIVE:

I. Estimate the complete response (CR) rate, time to response, duration of response (DOR), overall survival (OS) and event-free survival (EFS) in relapsed/refractory FL patients treated with tazemetostat, umbralisib and ublituximab.

EXPLORATORY OBJECTIVES:

I. Examine the immune effects of concurrent targeting of PI3K and EZH2 in patients with FL. II. Examine the evolution of tumor genetic profile while on therapy with tazemetostat, umbralisib and ublituximab, as determined by liquid biopsy.

OUTLINE: This is a phase I, dose-escalation study of tazemetostat and umbralisib followed by a phase II trials.

Patients receive ublituximab intravenously (IV) on days 1, 8, and 15 of cycle 1, day 1 of cycle 2-6, and day 1 of every 3 cycles thereafter. Patients also receive tazemetostat orally (PO) twice daily (BID) umbralisib by PO once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed diagnosis of follicular lymphoma grade 1-3a according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution
* Relapsed/ refractory disease after at least 2 lines of systemic therapy including an anti-CD20 antibody. Relapse must have been confirmed histologically (with hematopathology review at the participating institution). Exceptions may be granted with study PI approval
* Active disease meeting requiring treatment per treating physician's decision
* Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy with one or more sites of disease >= 1.5 cm in longest dimension
* Fully recovered from the acute toxic effects (except alopecia) to <= Grade 1 to prior anti-cancer therapy
* Without bone marrow involvement: Absolute neutrophil count (ANC) >=≥ 1,000/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement.
* With bone marrow involvement: ANC >= 500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement.
* Without bone marrow involvement: Platelets >= 50,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement.
* With bone marrow involvement: Platelets >= 30,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement.
* Hemoglobin >= 8 g/dL

  * NOTE: No erythropoietin and/or packed red blood cells (pRBC) transfusion allowed within 7 days prior to screening)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease or hepatic involvement by lymphoma)
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine clearance of >= 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* Women of childbearing potential (WOCBP): negative serum pregnancy test within 3 days prior to cycle 1 day 1
* Agreement by females of childbearing potential* to use 2 reliable methods of contraception simultaneously (including one highly effective and one effective contraceptive method) and males (including those who have had a vasectomy) to use an highly effective method of birth control, or abstain from heterosexual activity for the course of the study starting from at least 28 days prior to initiating tazemetostat for women, and 7 days prior to initiating tazemetostat for men, through at least 6 months after the last dose of tazemetostat for women and 3 months for men, and at least 4 months after the last dose of ublituximab or umbralisib, whichever comes later, for both men and women

  * Childbearing potential defined as not being surgically sterilized (women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Prior therapeutic intervention with any of the following: therapeutic anticancer antibodies within 3 weeks (rituximab); radio- or toxin-immunoconjugates within 10 weeks; all other chemotherapy or radiation therapy within 3 weeks prior to day 1 of protocol therapy.
* Prior exposure to either a PI3K inhibitor (including but not limited to idelalisib, duvelisib, copanlisib, and umbralisib) or an EZH2 inhibitor (including but not limited to tazemetostat).
* Prior allogeneic stem cell transplant
* Autologous hematologic stem cell transplant within 6 months of day 1 of protocol therapy
* Major surgical procedure (under general anesthesia) within 30 days of Day 1 of protocol therapy. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Chronic use of corticosteroids >= 20 mg/day of prednisone or equivalent (short-term use of steroids < 14 days is allowed).
* Requires treatment with a strong or moderate cytochrome P450 3A4 (CYP3A4) inhibitor/inducer
* Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components
* Concurrent participation in another therapeutic clinical trial
* History of prior malignancy. Exceptions include malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of protocol therapy; adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease; adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease; asymptomatic prostate cancer managed with "watch and wait" strategy.
* Prior history of myeloid malignancies including myelodysplastic syndrome (MDS) or presence of cytogenetic and/or molecular abnormalities known to be associated with MDS or myeloproliferative neoplasms (MPN) (e.g. del 5q, chr 7 abn, JAK2 V617). Any evidence of clonal hematopoiesis in the screening bone marrow biopsy should be discussed with the study principal investigator (PI) prior to enrollment
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass
* Known active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement
* Clinically significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class III or IV cardiac disease as defined by the New York Heart Association Functional Classification. Note Subjects with controlled, asymptomatic atrial fibrillation can enroll on study.
* Inability to swallow and retain an oral medication
* Clinically significant uncontrolled illness, including active infection requiring antibiotics
* Live virus vaccines within 4 weeks of start of protocol therapy or planned administration of live virus vaccines during ublituximab therapy
* Evidence of chronic active hepatitis B (HBV, not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody) or chronic active hepatitis C infection (HCV), or active cytomegalovirus (CMV). If hepatitis B virus core (HBc) antibody is positive, the subject must be evaluated for the presence of HBV deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR). If HCV antibody is positive, the subject must be evaluated for the presence of HCV ribonucleic acid (RNA) by PCR. If the subject is CMV IgG or CMV IgM positive, the subject must be evaluated for the presence of CMV DNA by PCR. Subjects with positive HBc antibody and negative HBV DNA by PCR are eligible. Subjects with positive HCV antibody and negative HCV RNA by PCR are eligible. Subjects who are CMV IgG or CMV IgM positive but who are CMV DNA negative by PCR are eligible. Patients with a prior known history of hepatitis B and those with a positive anti-HBc with negative hepatitis B surface antigen (HBsAg) at screening must be able to receive antiviral agents effective against hepatitis B such as, but not limited to, enofovir or entecavir
* Known history of human immunodeficiency virus (HIV) infection
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 28 days (1 cycle)
  Assessed by Common Terminology Criteria for Adverse Events version 5.0. Summarized by type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment, and reversibility or outcome.
Overall response rate | Up to 2 years
  Will be estimated by the proportion of response-evaluable patients achieving complete response (CR) or partial response (PR, along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Complete response rate | Up to 2 years
  Will be estimated by the proportion of response-evaluable patients achieving CR or PR, along with the 95% exact binomial confidence interval.
Time to response | Up to 2 years
  Will be summarized among those achieving CR/PR using descriptive statistics.
Duration of response | Up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Overall survival | From start of protocol treatment to time of death due to any cause, assessed up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Event-free survival | From start of protocol treatment to time of disease relapse/progression, start of non-protocol anti-lymphoma therapy due to toxicity of the protocol therapy, or death due to any cause, assessed up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mei, Principal Investigator — City of Hope Medical Center